CLINICAL TRIAL: NCT02793167
Title: Clinical Values of Automated Electronic Alert for Acute Kidney injury-a Prospective ,Randomly Controlled Cohort Study
Brief Title: Clinical Values of Automated Electronic Alert for Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XinLing Liang (Other)
Responsible Party: Sponsor-Investigator, XinLing Liang, Director of Blood Purification Center of Guangdong General Hospital, Guangdong Provincial People's Hospital
Organization: Guangdong Provincial People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: GGH2016-1
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; medication alert systems
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Usual care (No Intervention): patients will receive standard clinical care by the doctor in charge.
- AKI alert (Experimental): an AKI alert will send to the the doctor in charge.Our team of nephrologists would give suggestions if the doctor in charge issue consultation application.
  Interventions: Device: AKI alert

INTERVENTIONS:
Device: AKI alert
  Arms: AKI alert

SUMMARY:
Acute kidney injury (AKI) is common, serious and expensive.It is associated with significant mortality, morbidity and increased length of hospital stay.To improve clinical outcomes of AKI by early detection and timely referral to the renal,the investigators developed an electronic alert system which identifies all cases of AKI occurring in patients over 18 years.The system was also designed to collect data on AKI incidence one of the biggest tertiary hospital in China.

DETAILED DESCRIPTION:
A prospective, randomly controlled cohort study will be conducted agmong the patients with AKI who are detected by the use of AKI sniffer. The investigators chose to assess all inpatient serum creatinine results using a combination of "KDIGO" criteria.

The investigators randomly divided the patients into two groups:

1. Usual care : patients will receive standard clinical care by the primary physicians
2. AKI alert : an AKI alert will be sent to the the doctor in charge. Our team of kidney experts would give a suggestion if the the doctor in charge issue consultation applications.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with an Alert for AKI(based on KDIGO guidelines)

Exclusion Criteria:

* patients already on dialysis for AKI at the time of alert
* patients with End stage renal disease
* patients <18 years of age
* patients dissenting from participation according to the Ethics application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2016-03; Primary Completion 2021-12 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Adverse events during hospitalization | from start of AKI to discharge,up to 4 weeks
  cardiac shock/ need for intensive care/ cardiopulmonary resuscitation/ cardiac death/ death
Incidence of cardiovascular disease and its occurrence time followed up for 1 years | One year after discharge
  heart failure/ acute coronary syndrome/ readmission/cardiac readmission/ cardiovascular intervention or surgery
The AKI outcome and its occurrence time followed up for 1 years | One year after discharge
  AKI recovery/stop renal replacement therapy
AKI recovery/stop renal replacement therapy | from start of AKI to discharge,up to 4 weeks
  Glomerular filtration rate decreased/ new occurrence proteinuria/ original proteinuria aggravation

SECONDARY OUTCOMES:
Proportion of nephrology referral | from start of AKI to discharge,up to 4 weeks
Diagnostic rate of AKI at discharge | from start of AKI to discharge,up to 4 weeks
Follow-up rate after discharge | One year after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Dept,Guangdong General Hospital, Guangzhou, Guangdong, China